CLINICAL TRIAL: NCT05260944
Title: Power Lung Versus Acapella on Airway Clearance After Coronary Artery Bypass Graft Surgery
Brief Title: Power Lung Versus Acapella After Coronary Artery Bypass Graft Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Shymaa yussuf abo zaid, Assistant lecturer, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: P.T.REC/012/002682
Record Dates: First submitted 2022-02-08; First posted 2022-03-02 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Coronary Artery Bypass Graft Surgery

STUDY DESIGN:
Intervention Model Description: In the study three groups of patients will participated first, group A. Will receive acapella device.
  Second, group B. Will receive power lung device. Third, group C. Will receive only routine physical Therapy program.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The participants are the patients who undergoing coronary artery bypass graft surgery.
  The care providers are the cardiothoraci surgeon and the nursing staff. The investigator is the physical Therapy ( my self)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Group A. Thirty patients will receive a two supervised session using Acapella three sets for 10 repetitions two times daily from first day postoperative until 7 days, in addition to routine physiotherapy program (phase I cardiac rehabilitation, breathing exercises, postural drainage, Percussion and vibration).
  Interventions: Device: Acapella device
- Group B (Experimental): Thirty patients will receive a two supervised sessions using power lung device three sets for 10 repetitions from the first day postoperative until 7 days(André L.et al., 2016), in addition to routine physiotherapy program (phase I cardiac rehabilitation, breathing exercises, postural drainage, percussion and vibration).
  Interventions: Device: Power lung device
- Group C (Active Comparator): Thirty patients will receive only routine physical Therapy program.
  Interventions: Other: routine Physical Therapy program

INTERVENTIONS:
Device: Acapella device — patients will receive a two supervised sessions using acapella device three sets for 10 repetitions from the first day postoperative until 7 days, in addition to routine physiotherapy program (phase I cardiac rehabilitation, breathing exercises, postural drainage, percussion and vibration.
  Arms: Group A
Device: Power lung device — Group B. patients will receive a two supervised sessions using power lung device three sets for 10 repetitions from the first day postoperative until 7 days, in addition to routine physiotherapy program (phase I cardiac rehabilitation, breathing exercises, postural drainage, percussion and vibration.
  Arms: Group B
Other: routine Physical Therapy program — Group C. Thirty patients will receive only routine physical Therapy program
  Arms: Group C

SUMMARY:
The purpose of the study is to compare between the power lung versus acapella on airway clearance after coronary artery bypass graft surgery.

DETAILED DESCRIPTION:
In this part of the study the materials and methods will be presented under the following headings: subjects, equipments, procedures of the study and statistical procedures

1. Subjects. Ninty patients of both sexes will participate in this study with an age range of 40 to 50 years old. They will be chosen from outpatient clinic, Qena University Hospital.

   Patients will be randomely assigned into three groups:

   Group A: patients will receive a two supervised sessions using acapella device three sets for 10 repetitions from the first day postoperative until 7 days, in addition to routine physiotherapy program (phase I cardiac rehabilitation, breathing exercises, postural drainage, percussion and vibration.

   Group B: patients will receive a two supervised session using power lung device three sets for 10 repetitions two times daily from first day postoperative until 7 days, in addition to routine physiotherapy program (phase I cardiac rehabilitation, breathing exercises, postural drainage, Percussion and vibration).

   Group C. Patients will receive only routine physical Therapy program.
2. Equipment:

1. For evaluation: Arterial blood gases including: - paO2, paCO2, PH and O2 saturation. Spirometry measurements: - as forced vital capacity (FVC) andbforced expiratory volume in the first second (FEV1).

The incidence of PPCs and the length of postoperative stay: - using the Melbourne Group Scale Dyspnea. According to the revised or modified Borg scale or rating of perceived exersion.

The Rand SF 36 health survey questionnaire. 2. For treatment The power lung device. Acapella device.

ELIGIBILITY:
Inclusion Criteria:

* They will be from 40-50 years old.
* They will be patients undergo elective CABG surgery.
* Non productive cough postoperatively.
* Cough pain intensity > 5 as rated on a visual analogue scale (VAS) on postoperative day 1.

Exclusion Criteria:

* Patients with chronic chest diseases.
* Patients with an intensive postoperative care (ICU) stay > 48 hrs.
* Uncooperative patients.

Ages: 40 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-08-05 (Actual); Primary Completion 2023-07-05 (Estimated); Study Completion 2023-08-05 (Estimated)

PRIMARY OUTCOMES:
Arterial blood gases including: | One week
  Partial pressure of oxygen (paO2), partial pressure of carbon dioxide (paCO2), power of hydrogen (PH)and O2 saturation.

SECONDARY OUTCOMES:
Spirometry | One week
  As forced vital capacity (FVC), forced expiratory volume in the first second (FEV1) and the FEV1/FVC.

OTHER OUTCOMES:
Dyspnea | One week
  According to revised or modified Borg or rating of perceived exertion.
The incidence of postoperative pulmonary complications | One week
  According to Melbourne group scale.
Quality of life | One week
  According to the Rand SF 36 health survey questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Shymaa Y Abo zaid, Master, Principal Investigator — Assistant lecturer
Locations (1):
- Shymaa yussuf abo zaid, Qina, Egypt